CLINICAL TRIAL: NCT05455840
Title: A Prospective, Single-Center Investigation of the da Vinci SP® Surgical System in Anterior Mediastinal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101422A0
Record Dates: First submitted 2022-05-16; First posted 2022-07-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Robotic Surgical Procedure; Thymoma; Myasthenia Gravis
Keywords: single incision robotic minimal invasive surgery; robotic mediastinal tumor resection; da Vinci SP® surgical system
MeSH Terms: conditions — Thymoma; Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: thymothmectomy or extended thymectomy through Da Vinci SP platform
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Patients with qualified criteria will be enrolled in this study
  Interventions: Device: Da Vinci SP surgical platform

INTERVENTIONS:
Device: Da Vinci SP surgical platform — using Da Vinci SP platform in thymothymectomy or extended thymectomy

SUMMARY:
Endpoints (Outcome measures)：

1. Primary endpoint: Incidence of conversion rate during surgery

   - The primary performance endpoint will be assessed as the ability to successfully complete the planned mediastinal procedure with da Vinci SP System, with no conversion to open surgery, video-assisted thoracoscopic surgery (VATS), multi-port robotic surgery or approach requiring undocking of the da Vinci SP Surgical System in order to complete the planned procedure using the alternate approach. Use of additional assistant port(s) is not considered a conversion
2. Secondary endpoints: Incidence of treatment related adverse events - The safety endpoint will be assessed as the incidence of all intra-operative and post-operative adverse events that occur through the 30-day follow up period

DETAILED DESCRIPTION:
During the past several years, minimally invasive thoracic surgery has evolved from thoracoscopic approaches using 3 -4 ports to a single incision video-assisted thoracoscopic surgery (VATS) techniques. Recently, the experience acquired with the uniportal VATS technique through the intercostal space has allowed the development of a uniportal VATS subxiphoid or subcostal approach for anterior mediastinal tumor resections. The advantage of using a subxiphoid or subcostal entry is to reduce pain by avoiding possible trauma of intercostal nerves caused by thoracic incisions. However, the longer distance from the subxiphoid or subcostal incision to the anterior mediastinal area makes this approach more difficult to perform extended thymothymectomy. During this same period of evolution into uniportal VATS surgery, robotic thoracic surgery has gained popularity as an alternative to traditional VATS. The advantages of robotics are the ability to perform surgery more precisely with articulated or wristed instruments, motion scaling, and tremor filtration, as well as improved visualization thanks to 3D high-definition video. However, currently 4 -5 incisions are still necessary to perform anatomic robotic resections.Recently, there has been a convergence of these two trends-uniportal surgery and robotic-assisted surgery-and has resulted in a single port robotic system, the da Vinci SP by Intuitive Surgical Cooperation. For this new platform, investigators plan to practice in extended thymothymectomy

ELIGIBILITY:
Inclusion criteria

1. Age >20 and <75 years-old
2. Willing and able to provide informed consent
3. ASA≤ 3
4. The subject fulfills one or both of the following criteria:

   * Diagnosis of myasthenia gravis
   * Masaoka stage I or II thymoma; thymic mass ≤ 5 cm diameter
5. Class I-IV Myasthenia gravis according to the Myasthenia Gravis Foundation of America Scientific Session (MGFA)

Exclusion criteria. Myasthenia gravis or thymoma patients with

1. Congestive heart failure (NHYA > II)
2. Arrhythmia required medication control
3. Subjects with a known bleeding or clotting disorder
4. Subjects actively receiving therapeutic dose anticoagulation or anti-platelet medications at the time of operation
5. Subjects under immunomodulatory within 30 days prior to the planned surgery
6. Previous ipsilateral thoracic surgery or sternotomy
7. Uncontrolled illness 6 months prior to planned surgical procedure including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
8. Previous neoadjuvant medical and/or radiation therapy
9. Subject has a contraindication for general anesthesia or surgery
10. Uncontrolled myasthenia gravis symptoms at the time of scheduled surgery
11. Confirmed thymic carcinoma
12. Patients who are not suitable for performing endoscopic surgery.
13. Myasthenia gravis patients with positive serum MuSK antibody. -

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-04-11 (Estimated); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion rate | During Surgery
  The primary performance endpoint will be assessed as the ability to successfully complete the planned procedure with da Vinci SP System, with no conversion to thoracoscopic, multi-port robotic, or open surgery.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | One year
  The safety endpoint will be assessed as the incidence of all intra-operative and post-operative adverse events that occur through the 30-day follow up period. Rceord the Incidence of Treatment-Emergent Adverse Events in our recording form

CONTACTS AND LOCATIONS:
Overall Officials: Yin Kai Chao, MD,PHD, Principal Investigator — CHENG GUNG MEMORIAL HOSPITAL
Locations (1):
- Chang Gung Memeorial Hospital, Linkou Medical Center, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No